CLINICAL TRIAL: NCT04307290
Title: The Impact of Dexmedetomidine on Tourniquet Induced -Systemic Effects in Total Knee Arthroplasty Under Spinal Anesthesia-prospective Study.
Brief Title: Dexmedetomidine on Tourniquet Induced -Systemic Effects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee, Professor, M.D., Ph.D., Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WonkwangUH6
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Arthropathy of Knee; Spinal Anesthesia; Tourniquet; Ischemia-reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: dexmedetomidine (0.5 μg/kg bolus over 10 minutes, followed by 0.5 μg/kg/h infusion from 10 min before the start of surgery to the end of surgery), and CON group (n = 40) received an equivalent volume of normal saline bolus and infusion as placebo until the end of surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization sequence was created using Stata 9.0 (Stata Corp, College Station, TX, USA) statistical software and was stratified by center with a 1:1 allocation using random block sizes of 4. Assignments were concealed in sealed envelopes. Participants were randomly assigned following simple randomization procedures (computerized random numbers) to 1 of 2 treatment groups: DEX group (n = 40) received intravenous dexmedetomidine (0.5 μg/kg bolus over 10 minutes, followed by 0.5 μg/kg/h infusion from 10 min before the start of surgery to the end of surgery), and CON group (n = 40) received an equivalent volume of normal saline bolus and infusion as placebo until the end of surgery.
  Patients, attending anesthesiologists responsible for patient care, and nurses were all blinded to the anesthetic agent during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Experimental): received intravenous dexmedetomidine (0.5 μg/kg bolus over 10 minutes, followed by 0.5 μg/kg/h infusion from 10 min before the start of surgery to the end of surgery
  Interventions: Drug: Dexmedetomidine Hydrochloride, or Saline
- CON group (Placebo Comparator): received an equivalent volume of normal saline bolus and infusion as placebo until the end of surgery.
  Interventions: Drug: Dexmedetomidine Hydrochloride, or Saline

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride, or Saline — drug infusion from 10 min before the start of surgery to the end of surgery
  Other Names: precedex

SUMMARY:
Eighty patients were randomly assigned to either control (CON) or dexmedetomidine (DEX) group. DEX group received a loading dose of 0.5 µg/ kg of intravenous dexmedetomidine over 10 minutes, followed by a continuous infusion of 0.5 µg/kg/h until completion of the surgery. CON group received the same calculated volume of normal saline. Pain outcomes, metabolic and coagulative changes after tourniquet application, and after tourniquet release were investigated.

DETAILED DESCRIPTION:
A total of 80 patients aged between 20 and 80 years, American Society of Anesthesiologists (ASA) physical status class I-III, who were scheduled to undergo elective TKA were enrolled in this study. Patients with history of rheumatoid arthritis, diabetes mellitus, hepatic or renal disease, allergy to drug being studied, heart block greater than first degree, left ventricle ejection fraction < 55%, or chronic administration of anti-inflammatory drugs, or opioids were excluded. Patients with tourniquet times of less than 60 minutes or longer than 150 minutes or with conversion to general anesthesia during surgery were also excluded.

Randomization Randomization sequence was created using Stata 9.0 (Stata Corp, College Station, TX, USA) statistical software and was stratified by center with a 1:1 allocation using random block sizes of 4. Assignments were concealed in sealed envelopes. Participants were randomly assigned following simple randomization procedures (computerized random numbers) to 1 of 2 treatment groups: DEX group (n = 40) received intravenous dexmedetomidine (0.5 μg/kg bolus over 10 minutes, followed by 0.5 μg/kg/h infusion from 10 min before the start of surgery to the end of surgery), and CON group (n = 40) received an equivalent volume of normal saline bolus and infusion as placebo until the end of surgery.

Patients, attending anesthesiologists responsible for patient care, and nurses were all blinded to the anesthetic agent during the study period.

Anesthesia and perioperative care Standard monitoring included electrocardiography, noninvasive arterial blood pressure monitoring, and pulse oximetry. All patients received spinal anesthesia performed by an attending anesthesiologist and 500 mL Ringer's lactate solution was administered for hydration before spinal anesthesia.

Spinal anesthesia was performed in the lateral decubitus position with the operative knee uppermost. These patients received an intrathecal injection of 0.5% bupivacaine 15 mg in 5% glucose at the level of L4-5 via using a 25-gauge needle. Patients were then turned to the supine position and the level of sensory block evaluated by pinprick.

Peak level of sensory block, sensory dermatome at tourniquet pain, time between tourniquet application and onset of pain, and tourniquet pain were performed by an independent researcher at 5, 10, 15 and 20 min after the spinal injection and then at 10-minutes intervals until the complete resolution of the sensory block.

The affected extremity in all patients was exsanguinated with an Esmarch bandage, and a tourniquet was applied at a pressure of 300 mmHg during surgery.

When a poorly localized, diffuse pain is felt by the patient at variable times after tourniquet inflation, despite adequate sensory blockade during surgery, it was considered to be induced by the tourniquet if it was unrelated to the surgical field, described as tourniquet pain in the affected extremity. Supplemental analgesia with intravenous fentanyl 100 μg was to be administered if any patient experienced tourniquet pain at any time during the procedure. General anesthesia would be induced if intravenous fentanyl supplementation was insufficient. The need for supplemental intravenous fentanyl and any conversion to general anesthesia were recorded.

When intraoperative bleeding occurred, volume replacement with Ringer's lactate solution was managed according to the decision of an attending anesthesiologist instead of blood products.

Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP) and heart rate (HR) were monitored every five minutes until the end of surgery.

Hypotension was defined as a 30% reduction of basal MAP, which was treated with ephedrine 5 mg iv. When the HR was <50 beats/minute (bradycardia), glycopyrrolate 0.2 mg was administered intravenously.

Before the start of surgery, femoral nerve block to reduce postoperative pain were performed using a bolus of 20 mL of ropivacaine 0.75%. Concurrently, patient-controlled analgesia (PCA) pump containing fentanyl 1000 μg, ketorolac 150 mg, and ramosetron 0.6 mg in a total volume of 150 mL of saline was set to deliver a basal infusion of 2 mL/h and bolus doses of 1 mL, with a 15-min lockout period for postoperative analgesia. PCA volume consumed at 24 and 48 hours after surgery and total PCA volume consumed for 48 hr after surgery. Postoperative pain intensity at rest was measured using a 100 mm linear visual analog scale (VAS). The VAS score for pain at rest was measured at 24 and 48 hours after surgery.

Fentanyl 100 μg was administered for a pain VAS ≥ 50 or ketorolac 30 mg was given for a pain VAS < 50 or upon patient request.

Measurements of metabolic, coagulative and temperature changes. The arterial blood samples were obtained from a radial artery at 1 minute just before the start of spinal anesthesia as a baseline and at 10 min after tourniquet release.

5 mL of blood samples were extracted through radial artery and then 1 mL were collected in the heparinized syringe; following this, the remaining blood samples were immediately sent through the pneumatic tube system, guaranteeing their processing in the least amount of time possible, not greater than 5 minutes by institutional standards. The metabolic variables included pH, lactate, calcium, potassium, bicarbonate, CO2, base excess and coagulative change included antithrombin III activity.

Tympanic temperature measurements were made using Braun Thermoscan (Thermoscan Inc., San Diego, CA) inserted into the auditory canal at 1 minute just before the start of spinal anesthesia as a baseline and at 10 minutes after tourniquet release

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 20 and 80 years, American Society of Anesthesiologists (ASA) physical status class I-III, who were scheduled to undergo elective TKA

Exclusion Criteria:

* Patients with history of rheumatoid arthritis, diabetes mellitus, hepatic or renal disease, allergy to drug being studied, heart block greater than first degree, left ventricle ejection fraction < 55%, or chronic administration of anti-inflammatory drugs, or opioids were excluded. Patients with tourniquet times of less than 60 minutes or longer than 150 minutes or with conversion to general anesthesia during surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
total PCA volume consumed | for 48 hours after surgery
  patient-controlled analgesia (PCA) pump containing fentanyl 1000 μg, ketorolac 150 mg, and ramosetron 0.6 mg in a total volume of 150 mL of saline was set to deliver a basal infusion of 2 mL/h and bolus doses of 1 mL, with a 15-min lockout period for postoperative analgesia.

SECONDARY OUTCOMES:
hemodynamic variable | baseline, 10 min, 30 min, 60min after tourniquet application and 10 min after tourniquet release
  Systolic blood pressure ((mmHg)), diastolic blood pressure ((mmHg)), mean arterial blood pressure ((mmHg)) were monitored every five minutes until the end of surgery.
heart rate (hemodynamic variable) | baseline, 10 min, 30 min, 60min after tourniquet application and 10 min after tourniquet release
  heart rate (beats/min) was monitored every five minutes until the end of surgery.
Number of participants with metabolic variables | baseline, 10 min after tourniquet release
  5 mL of blood samples were extracted through radial artery and then 1 mL were collected in the heparinized syringe; following this, the remaining blood samples were immediately sent through the pneumatic tube system, guaranteeing their processing in the least amount of time possible, not greater than 5 minutes by institutional standards. The metabolic variables included pH, lactate(Mm/L), calcium(mg/dl), potassium(mEq/L), bicarbonate(Mm/L), CO2(mmHg)
coagulative variable | baseline, 10 min after tourniquet release
  coagulative change included antithrombin III activity (%).
body temperature | at 1 min just before the start of spinal anesthesia as a baseline and at 10 min after tourniquet release.
  Tympanic temperature measurements were made using Braun Thermoscan inserted into the auditory canal

CONTACTS AND LOCATIONS:
Locations (1):
- WonwangUH, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No